CLINICAL TRIAL: NCT02984969
Title: Characterization of Intestinal Microbiota in Constipation Patients: Using 16S rRNA Gene Sequencing Analysis
Brief Title: Using 16S rRNA Gene Sequencing Analysis Intestinal Microbiota in Constipation Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, PhD, Jinling Hospital, China
Other Study IDs: STC-2016-16sRNA
Record Dates: First submitted 2016-11-20; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Slow Transit Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Slow transit constipation: subjects met the Rome III criteria for STC
- Healthy subjects: Healthy controls

SUMMARY:
Constipation is a frequent, chronic gastroenterological problem that has many varied symptoms and thus has several clinical definitions. According to the Rome III criteria for chronic constipation, almost 16% of all adults are affected by chronic constipation worldwide, and it is more prevalent and symptomatic in women and elderly people. Slow transit constipation (STC) is the major category and is characterized by a decreased rate of colonic transit.

Recently, many researchers have focused on the relationship between intestinal microbiota and constipation and have demonstrated that intestinal microbiota contribute to the pathophysiology of functional gastrointestinal disorders.

Thus, there is a need for an improved understanding of gut microbiota composition in constipation patients and for the potential role played by the gut microbiota in the etiology of STC.To achieve this goal the investigators characterized and compared the intestinal microbiota among carefully selected patients with constipation that were clinically categorized based on Rome III criteria, and healthy controls using high throughput pyrosequencing of the 16S rRNA gene and a conservative approach to detect quantitative changes in the relative abundances of taxa.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic constipation according to Rome III criteria, defined as two or fewer spontaneous, complete bowel movements (SCBMs) per week for a minimum of 6 months;
2. Age > 18 years;
3. BMI: 18.5-25 kg/m2;
4. Slow colonic transit confirmed by colonic transit test (colonic transit time (CTT) > 48 hours);
5. Normal anorectal manometry, with no evidence of dyssynergia and confirmed ability to expel rectal balloon;
6. No radiographic evidence of functional (i.e. pelvic floor dyssynergia) or anatomical (i.e. significant rectocele and intussusception) impediment to the expulsion of the radio-opaque contrast;
7. Disease duration > 1 year;
8. Traditional treatment with dietary modification, laxatives (including osmotic and stimulant laxatives), and biofeedback tried over the past 6 months without success;

Exclusion Criteria:

1. Bowel constipation due to innate factor (i.e. megacolon) or secondary interventions (i.e. drugs, endocrine, metabolic, neurologic or psychologic disorders);
2. History or evidence of gastrointestinal diseases (i.e. obstruction, cancer, inflammatory bowel diseases) ;
3. Previous abdominal surgery, except cholecystectomy, appendicectomy, tubal ligation and cesarean section;
4. Previous proctological or perianal surgery;
5. A constipation condition meeting the Rome III criteria for IBS or functional abdominal pain syndrome;
6. Pregnant or breast-feeding women;
7. Infection with enteric pathogen;
8. Usage of probiotics, prebiotics and/or synbiotics within the last month;
9. Usage of antibiotics and/or PPIs within the last 3 months;
10. Smoking or alcohol addiction within the last 3 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 18 subjects met the Rome III criteria for STC and 17 healthy controls were recruit from Jinling Hospital, a teaching hospital of Nanjing University
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Fecal microbiota sequence | Within a week after enroll
  The fecal samples and isolated microbiota samples were frozen immediately and underwent DNA extraction using standard methods at BGI-Shenzhen

SECONDARY OUTCOMES:
Stool short-chain fatty acids (SCFAs) | Within a week after enroll
  The stool short-chain fatty acids (SCFAs) were extracted and quantitatively analysed by gas chromatography-mass spectrometry (GC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Tian, Principal Investigator — Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tian H, Chen Q, Yang B, Qin H, Li N. Analysis of Gut Microbiome and Metabolite Characteristics in Patients with Slow Transit Constipation. Dig Dis Sci. 2021 Sep;66(9):3026-3035. doi: 10.1007/s10620-020-06500-2. Epub 2020 Aug 7. PMID 32767153